CLINICAL TRIAL: NCT01494103
Title: Administration of Haploidentical Donor T Cells Transduced With the Inducible Caspase-9 Suicide Gene
Brief Title: Administration of Donor T Cells With the Caspase-9 Suicide Gene
Acronym: DOTTI
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Collaborators: The Methodist Hospital Research Institute (Other); Center for Cell and Gene Therapy, Baylor College of Medicine (Other)
Responsible Party: Principal Investigator, Malcolm Brenner, Director/Professor, Center for Cell and Gene Therapy, Baylor College of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H-28256-DOTTI; DOTTI (Other: Baylor College of Medicine)
Record Dates: First submitted 2011-12-15; First posted 2011-12-16 (Estimated); Last update posted 2025-07-11 (Actual); Status verified 2025-07

CONDITIONS: Acute Lymphoblastic Leukemia; Myelodysplastic Syndrome; Acute Myeloid Leukemia; Chronic Myelogenous Leukemia; Non Hodgkin Lymphoma; Hemophagocytic Lymphohistiocytosis; Familial Hemophagocytic Lymphohistiocytosis; Hemophagocytic Syndrome; Epstein Barr Virus Infection; X-linked Lymphoproliferative Disease
Keywords: Acute lymphoblastic leukemia; Myelodysplastic syndrome; Acute myeloid leukemia; Chronic myelogenous leukemia; Non Hodgkin lymphoma; Hemophagocytic lymphohistiocytosis; Familial hemophagocytic lymphohistiocytosis; Hemophagocytic syndrome; Epstein Barr virus infection; X-linked lymphoproliferative disease
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Myelodysplastic Syndromes; Leukemia, Myeloid, Acute; Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Lymphoma, Non-Hodgkin; Lymphohistiocytosis, Hemophagocytic; Epstein-Barr Virus Infections; Lymphoproliferative Disorders | interventions — AP 1903 reagent

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- iCaspase9-transduced T cells (Experimental): The 5 dose levels are:
  1. 1 x 10^4 T cells/kg
  2. 1 x 10^5 T cells/kg
  3. 5 x 10^5 T cells/kg
  4. 1 x 10^6 T cells/kg
  5. 5 x 10^6 T cells/kg
  AP1903 will be administered if there is development of Grade 1 or greater GvHD.
  Interventions: Biological: iCaspase9-transduced T cells; Drug: AP1903

INTERVENTIONS:
Biological: iCaspase9-transduced T cells — Patients will receive the T cells between 30 and 90 days following transplantation. The T cells will be infused through a catheter line.
Drug: AP1903 — AP1903 will be administered if there is development of Grade 1 or greater GvHD.
  Dose: 0.4 mg/kg by IV over 2 hours.
  Up to 3 additional doses may be administered if the GvHD does not respond or gets worse.
  Other Names: AP1903 Dimerizer Drug

SUMMARY:
Patients will be receiving a stem cell transplant as treatment for their disease. As part of the stem cell transplant, patients will be given very strong doses of chemotherapy, which will kill all their existing stem cells.

A close relative of the patient will be identified, whose stem cells are not a perfect match for the patient's, but can be used. This type of transplant is called "allogeneic", meaning that the cells are from a donor. With this type of donor who is not a perfect match, there is typically an increased risk of developing GvHD, and a longer delay in the recovery of the immune system.

GvHD is a serious and sometimes fatal side-effect of stem cell transplant. GvHD occurs when the new donor cells (graft) recognize that the body tissues of the patient (host) are different from those of the donor.

In this study, investigators are trying to see whether they can make special T cells in the laboratory that can be given to the patient to help their immune system recover faster. As a safety measure, we want to "program" the T cells so that if, after they have been given to the patient, they start to cause GvHD, we can destroy them ("suicide gene").

Investigators will obtain T cells from a donor, culture them in the laboratory, and then introduce the "suicide gene" which makes the cells sensitive to a specific drug called AP1903. If the specially modified T cells begin to cause GvHD, the investigators can kill the cells by administering AP1903 to the patient. We have had encouraging results in a previous study regarding the effective elimination of T cells causing GvHD, while sparing a sufficient number of T cells to fight infection and potentially cancer.

More specifically, T cells made to carry a gene called iCasp9 can be killed when they encounter the drug AP1903. To get the iCasp9 gene into T cells, we insert it using a virus called a retrovirus that has been made for this study. The AP1903 that will be used to "activate" the iCasp9 is an experimental drug that has been tested in a study in normal donors with no bad side-effects. We hope we can use this drug to kill the T cells.

The major purpose of this study is to find a safe and effective dose of "iCasp9" T cells that can be given to patients who receive an allogeneic stem cell transplant. Another important purpose of this study is to find out whether these special T cells can help the patient's immune system recover faster after the transplant than they would have otherwise.

DETAILED DESCRIPTION:
If the patient is doing well after the stem cell transplant, and does not have severe GvHD, s/he will be eligible to receive the special "iCasp9" T cells from Day 30 to 90 after transplant. The specially selected and treated T cells will be given by vein (IV) once.

This is a dose escalation study. This means that at the beginning, patients will be started on the lowest dose (1 of 5 different levels) of T cells. Once that dose schedule proves safe, the next group of patients will be started at a higher dose. This process will continue until all 5 dose levels are studied. If the side-effects are too severe, the dose will be lowered or the T cell injections will be stopped.

If the patient develops GvHD after being given the specially treated T cells, we will prescribe AP1903, which has been shown to kill cells carrying the iCasp9 gene. This drug will be given as a 2-hour IV infusion.

We will continue to follow the patient weekly in the bone marrow transplant clinic for the first month after the infusion, to check for side-effects of the treatment and for GvHD. The patient will have the standard tests performed that all patients have after transplant, even when not receiving special T cells.

ELIGIBILITY:
Inclusion Criteria:

Inclusion Criteria at Time of Procurement:

1. Lack of a suitable conventional donor (i.e. 5/6 or 6/6 related, or 5/6 or 6/6 unrelated donor), or presence of a rapidly progressive disease not permitting time to identify an unrelated donor.
2. High risk disease in one of the following:

   * Myelodysplastic syndrome (MDS) in one of the following categories: RCMD with an IPSS-R of intermediate, poor, or very poor, RAEB-1, or RAEB-2
   * Acute myeloid leukemia (AML) after first relapse or primary refractory disease
   * Chronic myelogenous leukemia (CML) in Chronic Phase 2 or greater, Accelerated Phase or Blast Crisis
   * Acute lymphoblastic leukemia (ALL) after first relapse or primary refractory disease, or High-Grade Non Hodgkin lymphoma (NHL) Stage III or IV after first relapse or primary refractory disease
   * Hemophagocytic lymphohistiocytosis (HLH)
   * Familial hemophagocytic lymphohistiocytosis (FLH)
   * Viral-associated hemophagocytic syndrome (VAHS)
   * T or NK cell lymphoproliferative syndrome
   * X-linked lymphoproliferative disease (XLP)

Inclusion Criteria at Time of T Cell Infusion:

1. Engrafted with an absolute neutrophil count (ANC) > 500 cells/µL
2. Greater than or equal to 50% donor chimerism in either peripheral blood or bone marrow, or relapse of their original disease
3. Life expectancy > 30 days
4. Lansky/Karnofsky score greater than or equal to 60
5. Absence of severe renal disease (creatinine > 2X upper limit of normal for age)
6. Absence of severe hepatic disease (direct bilirubin > 3X upper limit of normal or SGOT > 3X upper limit of normal)
7. Oxygen saturation > 94% on room air
8. Patient/Guardian able to give informed consent
9. AP1903 available in sufficient quantities to allow for treatment of the patient

Exclusion Criteria:

Exclusion Criteria at Time of T Cell Infusion:

1. GvHD
2. Severe intercurrent infection
3. Pregnancy*
4. Other investigational drugs in the prior 30 days

   * Pregnancy test only required for at-risk individuals, defined as female patients of childbearing potential who have received a reduced-intensity conditioning regimen.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2011-11; Primary Completion 2029-05 (Estimated); Study Completion 2029-05 (Estimated)

PRIMARY OUTCOMES:
Clinical and immunological effects of AP1903 administration. | 14 days
  To evaluate the clinical and immunological effects of AP1903 administration, a dimerizer drug used to activate an iCaspase9 suicide gene mechanism, to subjects who have received escalating doses of T lymphocytes expressing the iCaspase9 gene and developed acute graft-versus-host-disease (GvHD).

SECONDARY OUTCOMES:
T cell dose that produces a greater than 25% risk of Grade II or greater GvHD. | 42 days
  To discover the number of T cells/kg (up to 5 x 10^6/kg) that produce a greater than 25% risk of inducing Grade II or greater acute GvHD in these subjects.
Immune reconstitution and relative contribution of iCaspase9-modified T cells post-infusion. | Up to 15 years
  To measure the subsequent immune reconstitution of recipients of iCaspase9 modified T cells (and dimerizer drug), and assess the relative contribution of endogenous T cell recovery and infused gene-modified T cells.
Overall and disease-free survival. | 100 days and 1 year
  To measure the overall and disease-free survival of recipients of iCaspase9 T cells at 100 days and at 1 year post-transplant.

CONTACTS AND LOCATIONS:
Overall Officials: Malcolm K Brenner, MB, PhD, Principal Investigator — Baylor College of Medicine
Locations (2):
- United States (2):
  - Texas Children's Hospital, Houston, Texas
  - The Methodist Hospital, Houston, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zhou X, Dotti G, Krance RA, Martinez CA, Naik S, Kamble RT, Durett AG, Dakhova O, Savoldo B, Di Stasi A, Spencer DM, Lin YF, Liu H, Grilley BJ, Gee AP, Rooney CM, Heslop HE, Brenner MK. Inducible caspase-9 suicide gene controls adverse effects from alloreplete T cells after haploidentical stem cell transplantation. Blood. 2015 Jun 25;125(26):4103-13. doi: 10.1182/blood-2015-02-628354. Epub 2015 May 14. PMID 25977584